CLINICAL TRIAL: NCT01582828
Title: Serial Hybrid Atrial Fibrillation Ablation
Acronym: SHAFT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical problems
Sponsor: Medisch Spectrum Twente (Other)
Responsible Party: Principal Investigator, B. Oude Velthuis, Research fellow electrophysiology, Medisch Spectrum Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHAFT-01
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation
Keywords: atrial; fibrillation; pvi; vats; ablation; hybrid
MeSH Terms: conditions — Atrial Fibrillation | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epicardial (surgical) ablation (Active Comparator): Epicardial Pulmonary vein isolation
  Interventions: Procedure: Epicardial (surgical) ablation
- Hybrid (Experimental): Epicardial (surgical) ablation & Endocardial assessment
  Interventions: Procedure: Hybrid

INTERVENTIONS:
Procedure: Epicardial (surgical) ablation — * Pulmonary vein isolation with bipolar clamps and bipolar box lesion
  * Epicardial atrial appendage closure
  Arms: Epicardial (surgical) ablation
Procedure: Hybrid — Epicardial (surgical) ablation
  * Pulmonary vein isolation with bipolar clamps and bipolar box lesion
  * Epicardial atrial appendage closure
  Endocardial assessment after 6-8 weeks, checking for isolation and if necessary touch up by RF ablation
  Arms: Hybrid

SUMMARY:
Treatment of (long-standing) persistent atrial fibrillation (AF) remains cumbersome and the surgical (epicardial) approach seems to be the most effective. Still, however a significant amount of failures exist which is mostly due to incompleteness of the surgical ablation lines. Checking, and if necessary additional ablation, of these lines afterwards endocardially by the cardiologist (the so-called serial hybrid approach) could overcome this problem.

ELIGIBILITY:
Inclusion Criteria:

* patients are screened and accepted for pulmonary vein isolation according to the current guidelines
* long standing persistent or persistent AF as defined in the guidelines
* left atrial size needs to be more than >46 mm on long axis or >35 cc/m2
* CHADSVASC score should be more than 0 as an indicator of a substantial substrate for atrial fibrillation.

Exclusion Criteria:

* Significant coronary artery disease has to be excluded as a trigger for AF by means of cardiac CT, if necessary a coronary angiogram will be performed.
* Previous PVI ablation (epicardial or endocardial) or cardiac surgery.
* Significant valvular disease present on echo.
* Concomitant cardiac surgery needed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation Freedom | 12 months
  left sided atrial flutter and left atrial tachycardia

SECONDARY OUTCOMES:
re-isolation | 8-10 weeks
  number of pulmonary veins needing re-isolation by the EP
Percentage of cross-over | 1 year
  Percentage of cross-over from the surgical arm alone to surgery and serial hybrid ablation.
Complications | 1 year
  Number of complications and thrombo-embolic events in both groups
Atrial fibrillation Burden | 1 year
  Burden of AF in both groups if AF is still present.

CONTACTS AND LOCATIONS:
Overall Officials: Jurren van Opstal, MD PhD, Principal Investigator — Medisch Spectrum Twente
Locations (1):
- Medisch Spectrum Twente, Enschede, Overijssel, Netherlands